CLINICAL TRIAL: NCT01607268
Title: Proton Magnetic Resonance Spectroscopy in Primary Autonomic Failure
Brief Title: Magnetic Resonance Spectroscopy in Autonomic Failure
Status: Terminated | Type: Observational
Why Stopped: Could not enroll enough participants, and lost funding.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor and Associate Director Clinical Research Center, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 120574
Record Dates: First submitted 2012-05-17; First posted 2012-05-30 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pure Autonomic Failure; Multiple System Atrophy
Keywords: autonomic failure; mangenetic resonance; neurochemistry; neurotransmitter; glutamate
MeSH Terms: conditions — Pure Autonomic Failure; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pure Autonomic Failure: Pure autonomic failure is a type of primary autonomic failure characterized by peripheral autonomic nervous system impairment.
  Interventions: Procedure: Magnetic Resonance Spectroscopy Imaging
- Multiple System Atrophy: Multiple system atrophy is a type of primary autonomic failure characterized by central autonomic nervous system impairment.
  Interventions: Procedure: Magnetic Resonance Spectroscopy Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy Imaging — Proton magnetic resonance spectroscopy [1H-MRS] is an emerging imaging tool that allows for non-invasive assessment of brain neurochemistry in human subjects. This technique allows for in vivo quantification of the concentration of neurotransmitters and metabolites in discrete brain regions through detection of hydrogen nuclei in these molecules. Autonomic failure patients will undergo a single imaging session lasting 30 to 90 minutes (0.5-1.5 hours) in the Vanderbilt Human Imaging Institute.
  Other Names: MRS

SUMMARY:
This research study will be conducted in patients with primary autonomic failure, a disabling condition that is associated with low blood pressure upon standing. These patients are also not able to control for changes in their blood pressure due to a loss of cardiovascular reflexes that are mediated within the brain. The purpose of this study is to determine whether magnetic resonance spectroscopy (MRS), a non-invasive imaging technique, can measure levels of chemicals (neurotransmitters) in the dorsal medulla, a brain area important for control of cardiovascular function, in autonomic failure patients. Importantly, this study will determine whether there are differences in brain chemicals between patients with peripheral versus central origins of their autonomic failure. The hypothesis is that the neurotransmitter profile in the medulla will be intact in patients with peripheral autonomic failure compared to those with central impairment. Overall, this study will provide insight into understanding the mechanisms involved in autonomic failure and will determine whether a single session of MRS imaging can improve the ability to make an accurate diagnosis in these patients. This would lessen the need for more extensive and invasive clinical testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary autonomic failure who are already participating in the approved Vanderbilt study "Evaluation and Treatment of Autonomic Failure"
* Males and females of all races between 18 and 80 years of age
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnant women
* Patients with diagnosed Parkinson's Disease or secondary forms of autonomic failure
* Patients with severe claustrophobia
* Patients taking medications known to affect brain neurotransmitter levels [e.g., anti-depressants, barbiturates, benzodiazepines, gabapentin, namenda, sinemet]
* Patients with implanted medical devices [e.g., pacemakers, metal clips, cochlear implants, orthopedic hardware], lead-based tattoos or pieces of metal close to or in an important organ
* High-risk patients [e.g., heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction]
* Inability to give or withdraw informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol including significant abnormalities in clinical, mental, or laboratory testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary autonomic failure patients will be recruited from patients already in the hospital participating in the approved protocol "The Evaluation and Treatment of Autonomic Failure." Prospective participants come from several sources including clinic patients, former patients, referrals from other physicians, and subjects that read about the Autonomic Dysfunction Center on the Vanderbilt website.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
N-Acetylaspartate Levels | 0.5-1.5 hours
  Differences in levels of N-acetylaspartate in the dorsal medulla of pure autonomic failure versus multiple system atrophy patients using single session imaging.

SECONDARY OUTCOMES:
Myoinositol Levels | 0.5-1.5 hours
  Differences in levels of myoinositol in the dorsal medulla pure autonomic failure versus multiple system atrophy patients.
GABA Levels | 0.5-1.5 hours
  Differences in levels of the neurotransmitter GABA in the dorsal medulla of pure autonomic failure versus multiple system atrophy patients.
Creatinine Levels | 0.5-1.5 Hours
  Differences in levels of creatinine-containing compounds in the dorsal medulla of pure autonomic failure versus multiple system atrophy patients.
Choline Levels | 0.5-1.5 Hours
  Differences in levels of choline-containing compounds in the dorsal medulla of pure autonomic failure versus multiple system atrophy patients.
Glutamate Levels | 0.5-1.5 Hours
  Differences in levels of glutamate in the dorsal medulla of pure autonomic failure versus multiple system atrophy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States